CLINICAL TRIAL: NCT00000650
Title: An Assessment of the In Vivo Biological Effects of Diethyldithiocarbamate (DTC) in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Connaught Laboratories (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 166; 11141 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Evaluation; Ditiocarb; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Ditiocarb

INTERVENTIONS:
Drug: Ditiocarb sodium

SUMMARY:
To determine, in HIV-infected patients, the magnitude and duration of the biological effects of ditiocarb sodium (sodium diethyldithiocarbamate; DTC) that may be relevant to treatment of HIV infection.

DTC has been studied in previous clinical trials in HIV-infected patients with the suggestion of delay in disease progression to AIDS and improvement in CD4 counts while on the drug.

DETAILED DESCRIPTION:
DTC has been studied in previous clinical trials in HIV-infected patients with the suggestion of delay in disease progression to AIDS and improvement in CD4 counts while on the drug.

Two groups of patients, one group asymptomatic and the other with AIDS diagnosis, are enrolled in the study. All patients receive DTC intravenously once a week for two weeks. Drugs are given on days 1 and 8. Blood samples are drawn on days 1, 3, 5, 8, 10, and 12.

ELIGIBILITY:
Inclusion Criteria

Patients must:

* Have HIV infection.
* Be asymptomatic (group 1) or have AIDS (group 2).
* Be able to understand and follow instructions.

Concurrent Medication:

Allowed:

GROUP 2:

* Anti-HIV therapy.
* Systemic prophylaxis or maintenance therapy for any AIDS-defining opportunistic infection excluding agents considered immunomodulators or immunosuppressants.
* Topical nystatin.
* Clotrimazole troches.
* Acyclovir.
* Dapsone.
* Trimethoprim / sulfamethoxazole (T/S).
* Fluconazole.
* Ketoconazole.
* Aerosolized pentamidine.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

ALL PATIENTS:

* Known hypersensitivity to disulfiram or diethyldithiocarbamate (DTC).
* Transfusion dependence.

GROUP 1 PATIENTS ONLY:

* Oral candidiasis documented by morphology or by a response to antifungal therapy.
* Oral hairy leukoplakia.
* Occurrence of herpes zoster in a single dermatomal distribution.
* Recurrent seborrheic dermatitis.
* Unintentional weight loss in excess of 10 pounds or 10 percent of usual body weight within 2 years prior to study.
* Unexplained temperature above 38 degrees C on more than 5 consecutive days or on more than 10 days in any 30 days within 2 years of expected study entry.
* Unexplained diarrhea defined by two or more stools/day for at least 14 days during a 120-day interval.
* Evidence of clinically significant cardiac, respiratory, hepatic, gastrointestinal, endocrine, hematologic, psychiatric, neurologic, renal, or dermatologic disease as demonstrated by history, physical, and laboratory evaluation.

GROUP 2 PATIENTS ONLY:

* Concurrent neoplasms other than Kaposi's sarcoma or basal cell carcinoma of the skin.
* Diagnosis of an acute opportunistic infection within 3 weeks of study entry or had treatment initiated for an opportunistic infection within 3 weeks of study entry.

Concurrent Medication:

Excluded:

ALL PATIENTS:

* Recombinant erythropoietin.

GROUP 1:

* Antiretroviral medications.

GROUP 2:

* Immunomodulators or immunosuppressants.

Concurrent Treatment:

Excluded:

* Requirement for blood transfusions more than once a month.

Patients with the following prior conditions are excluded:

GROUP 1 PATIENTS ONLY:

* Oral candidiasis documented by morphology or by a response to antifungal therapy.
* Oral hairy leukoplakia.
* Occurrence of herpes zoster in a single dermatomal distribution.
* Recurrent seborrheic dermatitis.
* Unintentional weight loss in excess of 10 pounds or 10 percent of usual body weight within 2 years prior to study.
* Unexplained temperature above 38 degrees C on more than 5 consecutive days or on more than 10 days in any 30-day period within 2 years of expected study entry.
* Unexplained diarrhea defined by two or more stools/day for at least 14 days during a 120-day interval.
* Evidence of clinically significant cardiac, respiratory, hepatic, gastrointestinal, endocrine, hematologic, psychiatric, neurologic, renal, or dermatologic disease as demonstrated by history, physical, and laboratory evaluation.

GROUP 2 PATIENTS ONLY:

* Diagnosis of an acute opportunistic infection within 3 weeks of study entry or had treatment initiated for an opportunistic infection within 3 weeks of study entry.

Prior Medication:

Excluded:

ALL PATIENTS:

* Corticosteroids, cytotoxic agents, or immunomodulating agents within 30 days prior to study entry.
* Chronic Antabuse (disulfiram) therapy.

GROUP 1 ONLY:

* Antiretrovial medications within 1 week prior to study entry.

Prior Treatment:

Excluded:

* Transfusion within 7 days of study entry.
* Radiation therapy within 30 days prior to study entry.

Unable to refrain from the use of alcohol for the duration of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12
Dates: Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PS Lietman, Study Chair; P Barditch-Crovo, Study Chair
Locations (1):
- Johns Hopkins Adult AIDS CRS, Baltimore, Maryland, United States